CLINICAL TRIAL: NCT00475592
Title: Validation of Esophageal Variceal Grading: A Comparative Study of Upper Gastrointestinal (GI) Endoscopy and Capsule Endoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study failed to recruit
Sponsor: Johns Hopkins University (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VaricealGrading_EsoCapsule
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Esophageal and Gastric Varices
Keywords: Esophageal Varices; Gastric Varices; Capsule Endoscopy; Portal Hypertension; Cirrhosis; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Esophageal and Gastric Varices; Hypertension, Portal; Fibrosis; Gastrointestinal Hemorrhage | interventions — Endoscopy; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capsule Endoscopy (Experimental)
  Interventions: Device: Esophageal Capsule Endoscopy
- Upper Gastrointestinal Endoscopy (Active Comparator)
  Interventions: Device: Upper Gastrointestinal Endoscopy

INTERVENTIONS:
Device: Esophageal Capsule Endoscopy
  Arms: Capsule Endoscopy
Device: Upper Gastrointestinal Endoscopy
  Arms: Upper Gastrointestinal Endoscopy

SUMMARY:
The purpose of this study is to develop a grading system for esophageal varices using capsule endoscopy in patients with portal hypertension and cirrhosis.

DETAILED DESCRIPTION:
Up to 35% of patients with cirrhosis will develop esophageal varices, which carry with them a 1-year and 3-year bleeding rate of 33% and 41%, respectively. Screening for varices with a video endoscopy is limited by its cost, patient compliance, and the risks of sedating a patient with portal hypertension. Capsule endoscopy is a novel method that may reduce the costs and increase compliance for screening.

The investigators propose to screen 100 consecutive patients with advanced cirrhosis for esophageal varices. A capsule endoscopy and video endoscopy will be done on the same day. The varices seen on video endoscopy will be graded using a standard grading scale. Both capsule and video endoscopy images will be assessed in a blinded fashion by 4 independent investigators. Finally, the video endoscopic images will be compared to capsule endoscopy to develop a capsule endoscopy grading system that corresponds to video endoscopy.

The primary endpoint of the study will be to develop a grading system for esophageal varices using capsule endoscopy. Secondary endpoints of the study include sensitivity, specificity, inter- and intraobserver variation of variceal grading using capsule endoscopy; patient acceptance as assessed on a visual analogue scale; and a cost comparison (facility fees + professional fees) of the two screening methods.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cirrhosis with portal hypertension based on imaging, clinical suspicion, or liver biopsy
* Age greater than or equal to 18 years old
* Able to give consent

Exclusion Criteria:

* Current implantable cardioverter-defibrillators or pacemaker in place
* Suspected intestinal obstruction
* Esophageal swallowing disorder
* Esophageal stenosis
* Age less than 18 years old
* Pregnancy
* Known Zenker's diverticulum
* Patients with previous endoscopic or surgical esophageal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be to develop a grading system for esophageal varices using capsule endoscopy. | Two years

SECONDARY OUTCOMES:
Secondary endpoints include sensitivity, specificity, inter- and intraobserver variation of variceal grading using capsule endoscopy; patient acceptance; and a cost comparison (facility + professional fees) of the two screening methods. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Thuluvath, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States